CLINICAL TRIAL: NCT03262259
Title: Measurement and Evaluation of Global Smart Drinking Goals Initiative
Brief Title: Evaluation of Global Smart Drinking Goals Initiative
Acronym: GSDG
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: HBSA (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0881
Record Dates: First submitted 2017-08-21; First posted 2017-08-25 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Binge Drinking, Underage Drinking, Drinking and Driving, Alcohol-Related Harms
MeSH Terms: conditions — Binge Drinking; Underage Drinking

STUDY DESIGN:
Intervention Model Description: Nine pairs of intervention and comparison cities followed over multiple years.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GSDG Intervention (Experimental): Cities receiving a multi-component intervention, including screening and brief intervention, other evidence-based interventions (e.g., enforcement of drink-driving or underage drinking laws), and novel or partially tested interventions that warrant further evaluation.
  Interventions: Behavioral: GSDG multi-component intervention
- Comparison (No Intervention): Comparison cities receiving no evidence-based interventions.

INTERVENTIONS:
Behavioral: GSDG multi-component intervention — Multi-component intervention, including screening and brief intervention, other evidence-based interventions, and novel or partially tested interventions that warrant further evaluation.
  Arms: GSDG Intervention

SUMMARY:
This study will evaluate effects of a multi-component, population-level intervention on alcohol use and related harms in six intervention cities relative to six matched comparison cities. Intervention components include screening and brief interventions by health providers, other evidence-based interventions (e.g., enforcement of drink-driving or underage drinking laws), and novel or partially tested interventions that warrant further evaluation. Key outcomes of interest include alcohol-related harms such as alcohol-related motor vehicle crashes and fatalities, heavy/binge drinking, underage drinking, and drinking and driving.

DETAILED DESCRIPTION:
This study will evaluate effects of a multi-component, population-level intervention on alcohol use and related harms in six intervention cities relative to six matched comparison cities. The trial is expected to expand to nine intervention and nine comparison cities in 2018. Intervention components include screening and brief interventions by health providers, other evidence-based interventions (e.g., enforcement of drink-driving or underage drinking laws), and novel or partially tested interventions that warrant further evaluation. Key outcomes of interest include alcohol-related harms such as alcohol-related motor vehicle crashes and fatalities, heavy/binge drinking, underage drinking, and drinking and driving.

Multiple years of pre- and post-intervention survey data will be collected from cross-sectional samples of adults and youth in each city to assess intervention effects on harmful alcohol use. Multiple years of archival data will also be collected from each city to assess intervention effects on alcohol-related harms such as motor vehicle crashes and fatalities, violence and unintentional injuries. Multi-level analyses will be conducted with data for the total sample of 18 cities and for each pair of cities to determine whether the overall goal of reducing harmful alcohol use by at least 10% is achieved.

ELIGIBILITY:
Inclusion Criteria:

* At least 12 years old
* Parental consent is be required if under 18 years old

Exclusion Criteria:

* Institutionalized individuals

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 36000 (Estimated)
Dates: Start 2017-09-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Health and social harms related to alcohol use | 1 year
  Self-reported problems related to alcohol use (e.g., drinking and driving, injury, unwanted sex, vandalism, property crime); alcohol-related motor vehicle crashes and fatalities

SECONDARY OUTCOMES:
Heavy/binge drinking | 1 year
  Self-reported heavy alcohol use (e.g., 5+ drinks within 2 hours)
Underage drinking | 1 year
  Self-reported alcohol use
Perceived alcohol use and alcohol-related attitudes among family and friends | 1 year
  Beliefs regarding alcohol use among family and friends, and acceptability of alcohol use
Alcohol expectancies | 1 year
  Expectations regarding positive and negative consequences of alcohol use
Awareness of alcohol policies | 1 year
  Knowledge of policies such as the minimum legal drinking age and maximum allowable blood alcohol concentration limit for driving
Perceived enforcement of alcohol policies | 1 year
  Perceived likelihood of being asked for age identification, being stopped by police for drinking and driving, etc.
Awareness of chronic health risks associated with alcohol use | 1 year
  Self-reported knowledge of possible chronic health-related consequences of alcohol use (e.g., liver cirrhosis, coronary heart disease)
Awareness of alcohol health guidance labels and information | 1 year
  Self-reported knowledge of guidance labels and information on beer bottles, cans and elsewhere
Consumption of no-alcohol and low-alcohol beer | 1 year
  Self-reported consumption (quantity and frequency) of no-alcohol and low-alcohol beer, no-alcohol and low-alcohol beer sales, underage use of no-alcohol and low-alcohol beer
Screening and brief intervention for heavy/binge drinking | 1 year
  Self-reported frequency and impacts, archival medical record data

CONTACTS AND LOCATIONS:
Overall Officials: Ted Miller, Ph.D., Principal Investigator — HBSA
Locations (1):
- HBSA, Calverton, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified survey and archival data collected for the evaluation will be made available upon completion of the study.
Supporting Information: Study Protocol
Time Frame: Data will become available upon completion of the study for an indefinite period.
Access Criteria: Not yet available.